CLINICAL TRIAL: NCT06993077
Title: Association Between Ultraviolet Radiation, Environmental Factors, and Ocular Biomechanical Properties: A Multicenter Cross-Sectional Study
Brief Title: Impact of Ultraviolet Radiation and Environmental Factors on Human Ocular Biomechanics
Status: Active, not recruiting | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2025010
Record Dates: First submitted 2025-04-15; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: environment Exposure — No special intervention

SUMMARY:
This observational study aims to explore whether ultraviolet (UV) radiation and other environmental factors are associated with ocular biomechanical properties in healthy volunteers aged 18-44 years without ocular diseases, ocular surgery history, or systemic diseases.

The main questions it aims to answer are:

Is there a significant correlation between UV radiation levels and corneal biomechanical parameters?

Do environmental factors such as geographic region and seasonal variation affect corneal biomechanical behavior?

Researchers will compare ocular biomechanical parameters among populations from different geographic regions with varying levels of UV radiation to determine whether there are statistically significant correlations or differences.

Participants will:

Undergo standardized ophthalmic examinations, including visual acuity, intraocular pressure, slit-lamp evaluation, axial length, and corneal topography;

Receive corneal biomechanical assessments using the Corvis ST device;

Provide basic demographic information and medical history;

Have all data de-identified, with the study strictly following ethical approval and privacy protection protocols.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

Age between 18 and 44 years (based on WHO criteria);

Spherical equivalent refraction (SER) ≤ 6.00 diopters;

No other ocular diseases;

No systemic diseases (e.g., diabetes, hypertension, cardiovascular diseases);

No severe psychiatric or psychological disorders;

No history of ocular surgery.

Exclusion Criteria

Severe psychiatric disorders;

Individuals diagnosed with keratoconus, suspected keratoconus, or subclinical keratoconus (based on the Global Consensus on Keratoconus Diagnosis);

Presence of other ocular diseases (e.g., glaucoma, corneal opacity, uveitis);

History of intraocular or ocular surface surgeries;

Presence of nystagmus or inability to cooperate with examinations;

History of intraocular surgery;

Presence of systemic diseases (e.g., diabetes, hypertension, cardiovascular diseases).

Exclusion Criteria:

* Severe psychiatric disorders;

Individuals diagnosed with keratoconus, suspected keratoconus, or subclinical keratoconus (based on the Global Consensus on Keratoconus Diagnosis);

Presence of other ocular diseases (e.g., glaucoma, corneal opacity, uveitis);

History of intraocular or ocular surface surgeries;

Presence of nystagmus or inability to cooperate with examinations;

History of intraocular surgery;

Presence of systemic diseases (e.g., diabetes, hypertension, cardiovascular diseases).

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will include individuals aged 18 to 44 years who are undergoing routine ophthalmic examinations across multiple medical centers. Participants must have no history of ocular or systemic diseases and meet specific refractive criteria. Only one eye per subject will be analyzed, and all biomechanical measurements will be performed using the same model of Corvis ST device to ensure consistency.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Corneal Biomechanical Parameters Measured by Corvis ST | Baseline (at time of examination)
  Central corneal thickness (CCT) mm
Corneal Biomechanical Parameters Measured by Corvis ST | Baseline (at time of examination)
  ,biomechanically corrected intraocular pressure (bIOP) mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, China, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided